CLINICAL TRIAL: NCT04210141
Title: An Adaptive Clinical Trial to Determine the Optimal Initial Dose of Lyophilized, Species Specific Monovalent Antivenom for the Management of Systemic Envenoming by Daboia Siamensis (Eastern Russell's Viper) in Myanmar
Brief Title: Optimal Dose of Antivenom for Daboia Siamensis Envenomings
Acronym: ODADS
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: due to current political circumstances in study site area.
Sponsor: Myanmar Oxford Clinical Research Unit (Other)
Collaborators: University of Oxford (Other); Mahidol Oxford Tropical Medicine Research Unit (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OXTREC 63-19
Record Dates: First submitted 2019-12-20; First posted 2019-12-24 (Actual); Last update posted 2024-04-01 (Actual); Status verified 2023-10

CONDITIONS: Daboia Siamensis Envenoming

STUDY DESIGN:
Intervention Model Description: Randomized adaptive design
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care (Active Comparator): Patients will receive an initial antivenom dose of 80mL lyophilized BPI viper antivenom, as per current national guidelines
  Interventions: Biological: lyophilized BPI viper antivenom
- Adaptive arm (Experimental): Patients will receive an initial dose of lyophilized BPI viper antivenom determined by the adaptive model.
  Interventions: Biological: lyophilized BPI viper antivenom

INTERVENTIONS:
Biological: lyophilized BPI viper antivenom — Antivenom

SUMMARY:
The aim of the study is to identify an 'optimal' initial dosing of the new Burma Pharmaceutical Industry (BPI) lyophilized mono-specific antivenom for patients with systemic Daboia siamensis envenoming. The initial dosing will aim to reverse venom-induced coagulopathy (as demonstrated by a negative 20 minutes Whole Blood Clotting Time (20WBCT) at 6 hours in 95% of patients whilst causing less than 5% anaphylactic reaction.

DETAILED DESCRIPTION:
Snake-bite envenoming (SBE) was re-categorized as a priority neglected tropical disease by the World Health Organization (WHO) in 2017. Antivenom is considered to be one of the most cost effective health interventions. Despite this, due to challenges in manufacture, reliance on cold chain for transport and storage, and geographically remote location of most envenomed patients, many patients do not receive the antivenom they require in a timely manner. The WHO strategy for a globally coordinated response to SBE highlighted the need to prioritize clinical research into the safety and effectiveness of antivenoms.

Myanmar is a country with a high incidence of snake-bite with an estimated 25,000 snake-bites and 1250 deaths per year. Daboia siamensis (Eastern Russell's viper) is responsible for 85% of snake-bites presenting to hospitals in Myanmar. Given their natural habitat and abundance of prey within the paddy fields, envenoming predominantly occurs in rural areas affecting agricultural workers.

Following a recent 4-year collaborative initiative between institutions in Myanmar and Australia entitled the Myanmar Snakebite project, antivenom production facilities have improved resulting in the production of a new monospecific lyophilized F(ab)'2 antivenom (Viper antivenom BPI). The new lyophilized antivenom has replaced the former liquid antivenom and has been distributed countrywide. The current dosing strategy is based on unpublished results of pre-clinical testing and stratified into two doses according to absence or presence of clinical features of severity at presentation (80 mL and 160 mL, respectively). No clinical trial data or post marketing data has been published to support the efficacy or toxicity of these recommended doses. This lack of robust clinical evidence to support dosing of antivenom is mirrored across the world with few well conducted trials to determine the safety and efficacy of antivenoms.

This paper presents a novel phase 2, model based, Bayesian adaptive design to determine optimal antivenom dosing for Russell's viper envenoming. In this context there are two concurrent considerations for dose optimality. Firstly, the efficacy of the dose, defined in this context as restoration of blood coagulation within 6 hours; secondly, the dose-related toxicity, defined as the occurrence of an anaphylactic reaction within 180 minutes post antivenom administration. The model based design estimates dose-response curves for both the efficacy outcome and the toxicity outcome, and thus derives a user-defined 'optimal dose'. Patients will be randomized at a ratio of 4:1 to either adaptive dose or standard of care respectively.

The study team will perform a number of nested studies within the dose finding trial:

* An assessment of the pharmacokinetic properties of Daboia siamensis venom pre and post antivenom administration.
* A parallel observation study of severely envenomed patients who will be administered 160mL (current standard of care).
* Sensitivity and specificity analysis of the 20WBCT and point of care International Normalized Ratio at detecting coagulopathy.
* A prospective follow up of envenomed patients to define the envenoming sequelae of Daboia siamensis envenoming.
* An assessment of ferryl-haem derivatives in urine of envenomed patients.

ELIGIBILITY:
Inclusion Criteria:

1. Patients suspected of systemic envenoming with DS
2. Incoagulable blood by 20-minute WBCT
3. Antivenom naïve
4. Age ≥ 15

Exclusion Criteria:

1. Receiving anticoagulant therapy e.g. warfarin
2. Known bleeding disorder e.g. haemophilia
3. Decompensated liver disease
4. Severely envenomed patients (as defined in the Myanmar National Guidelines)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-04 (Estimated); Primary Completion 2027-02-01 (Estimated); Study Completion 2027-11-01 (Estimated)

PRIMARY OUTCOMES:
Blood Coagulation | within 24 hours of patient recruitment
  Blood coagulation at 6 hours as measured by the 20 minute WBCT (binary outcome)
Anaphylaxis | within 24 hours of patient recruitment
  Anaphylaxis as defined by the European Academy of Allergy and Immunology within 180 minutes of antivenom administration

SECONDARY OUTCOMES:
Time to restoration of blood coagulability as determined by the 20 WBCT. | within 24 hours of patient recruitment
International normalized ratio (INR) determined by the POC INR meter. | within 24 hours of patient recruitment
Blood coagulability as determined by PT and fibrinogen | within 24 hours of patient recruitment
Occurrence of any serious adverse events | within 24 hours of patient recruitment
The occurrence of envenoming sequelae at 3 month follow up | within 6 months of patient recruitment
The occurrence of detectable ferryl-haem derivatives in urine samples | within 6 months of patient recruitment
The occurrence of Capillary Leak Syndrome | within 2 weeks of patient recruitment

CONTACTS AND LOCATIONS:
Locations (1):
- Myanmar Oxford Clinical Research Unit, Yangon, Burma

IPD SHARING:
Plan to Share IPD: Undecided
For ethics purposes, there is no current plans to share IPD with other researchers.

REFERENCES:
- [Background] Gutierrez JM, Calvete JJ, Habib AG, Harrison RA, Williams DJ, Warrell DA. Snakebite envenoming. Nat Rev Dis Primers. 2017 Sep 14;3:17063. doi: 10.1038/nrdp.2017.63. PMID 28905944
- [Background] Williams DJ, Faiz MA, Abela-Ridder B, Ainsworth S, Bulfone TC, Nickerson AD, Habib AG, Junghanss T, Fan HW, Turner M, Harrison RA, Warrell DA. Strategy for a globally coordinated response to a priority neglected tropical disease: Snakebite envenoming. PLoS Negl Trop Dis. 2019 Feb 21;13(2):e0007059. doi: 10.1371/journal.pntd.0007059. eCollection 2019 Feb. No abstract available. PMID 30789906
- [Background] Myint-Lwin, Warrell DA, Phillips RE, Tin-Nu-Swe, Tun-Pe, Maung-Maung-Lay. Bites by Russell's viper (Vipera russelli siamensis) in Burma: haemostatic, vascular, and renal disturbances and response to treatment. Lancet. 1985 Dec 7;2(8467):1259-64. doi: 10.1016/s0140-6736(85)91550-8. PMID 2866333
- [Background] Alfred S, Bates D, White J, Mahmood MA, Warrell DA, Thwin KT, Thein MM, Sint San SS, Myint YL, Swe HK, Kyaw KM, Zaw A, Peh CA. Acute Kidney Injury Following Eastern Russell's Viper (Daboia siamensis) Snakebite in Myanmar. Kidney Int Rep. 2019 May 29;4(9):1337-1341. doi: 10.1016/j.ekir.2019.05.017. eCollection 2019 Sep. No abstract available. PMID 31517153
- [Background] Wheeler GM, Mander AP, Bedding A, Brock K, Cornelius V, Grieve AP, Jaki T, Love SB, Odondi L, Weir CJ, Yap C, Bond SJ. How to design a dose-finding study using the continual reassessment method. BMC Med Res Methodol. 2019 Jan 18;19(1):18. doi: 10.1186/s12874-018-0638-z. PMID 30658575